CLINICAL TRIAL: NCT02714426
Title: A 14 Week Study of Mindfulness Effects on Attentional Control in Older Adults (The MACS Study: Mindfulness and Attentional Control in Seniors)
Brief Title: A 14 Week Study of Mindfulness Effects on Attentional Control in Older Adults
Acronym: MACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB02-2016-U-0277-N; 1F31AG051356-01A1 (NIH); IRB201800586 (Other: UF IRB)
Record Dates: First submitted 2016-03-10; First posted 2016-03-21 (Estimated); Results first posted 2019-02-21 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-02

CONDITIONS: Cognitive Aging
Keywords: Cognitive Aging; Attention; Mindfulness
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain Health (Active Comparator): In weeks 1 and 14, participants receive: Montreal Cognitive Assessment (MoCA), Wechsler Test of Adult Reading (WTAR), Functional Activities Questionnaire (FAQ), Older Americans Resources and Services (OARS) Complete Activities of Daily Living Scale, The Short Form (36) Health Survey (SF-36), Attention measures (Attention Network Test (ANT); Continuous Performance Test (CPT); Auditory Dual Task (ADT); Mind wandering; Cued Stroop), Positive and Negative Affect Scale (PANAS), Geriatric Depression Scale (GDS), Mindfulness Attention Awareness Scale (MAAS), Five Facet Mindfulness Questionnaire (FFMQ), Emotion Regulation Questionnaire (ERQ), State-Trait Anxiety Inventory (STAI), and Starkstein Apathy Scale (AS). In weeks 4-11, participants receive the Brain Health control instruction.
  Interventions: Other: Brain health
- Mindfulness-inspired Treatment/Testing (Experimental): Participants receive all of the same measures as the active comparator "Brain Health" condition in Weeks 1-14. In weeks 4-11, participants receive Mindfulness Inspired Treatment
  Interventions: Behavioral: Mindfulness-inspired treatment

INTERVENTIONS:
Behavioral: Mindfulness-inspired treatment — Eight weekly group MIT sessions lasting 90-120 minutes, along with a ½ day Mindfulness Retreat at the end of the training period, will include 1) psychoeducation, 2) formal exercises in the form of guided practice mentioned above, and 3) thoughtful exploration of ideas and questions. Formal MIT training will follow 21 guided pre-recorded meditative Moving Picture Experts Group Layer-3 Audio (MP3) tracks from the authors for use in class and at home, promoting both fidelity to the model and uniformity in intervention across training groups. MIT activities in the protocol include mindful breathing, eating, walking, and various other practices well documented in the literature to promote mindfulness. Participants will be asked to practice MIT on their own time, and to log this.
  Other Names: Mindfulness-based stress reduction
  Arms: Mindfulness-inspired Treatment/Testing
Other: Brain health — Eight weekly group brain health sessions lasting 90-120 minutes. The intervention is psychoeducational, and each week presents information from NIH regarding factors that may promote cognitive health in late life (e.g., sleep, physical activity, social engagement and leisure, cognitive training). Weekly sessions are supplemented with educational videos and group discussion. Weekly homework consists of readings about brain health.
  Other Names: Active comparator
  Arms: Brain Health

SUMMARY:
Attentional control, or individuals' ability to choose which stimuli in the environment they attend to and which they ignore, declines with older age. Studies from the past two decades suggest that mindfulness meditative practice, such as a standardized mindfulness based stress reduction programs, may increase the efficiency of attention networks.To date, the majority of studies that have related mindfulness meditation practice to attentional control have been based on retrospective self-reported mindfulness or cross-sectional measurement in experienced meditators. More recent experimental studies using pre-post training designs have shown that meditation-naïve individuals can experience attentional improvement with mindfulness intervention. This study seeks to elucidate the time course and process by which such attentional improvements might be achieved.

This research study investigates change in attentional control as participants progress through an 8-week mindfulness-inspired training (MIT) intervention, and has two specific aims: 1) to determine the time course of change in attentional components such as cognitive control and sustained attention as a consequence of MIT; attention will be measured weekly for 3 weeks before, 3 weeks after, and during 8 weeks of MIT. 2) To investigate the extent to which change in attentional performance is coupled/correlated with markers of emotion regulation, perceived mindfulness, and perceived mind wandering.

DETAILED DESCRIPTION:
This will be a 14-week research study exploring week to week changes in attentional control and selected time-varying covariates. The study will involve comparison of two groups of adults aged 65 and older. Half the participants (n=20) will be randomized to received eight weeks of mindfulness-inspired training, while the other half (n=20) are not.

Groups will be compared in the amount of change experienced in measures of attentional control. In addition, the association between changes in emotion regulation, perceived mindfulness, and perceived mind wandering with changes in attentional control will be examined, as well as whether this association differs between persons who did and did not receive mindfulness-inspired training. Measurement will include both paper-and-pencil and computer-administered tests.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent and perform cognitive and behavioral (mindfulness) interventions;
* Time and willingness to commit to the completion of this study;
* Ability to read at an 8th grade level based on scores on the Wechsler Test of Adult Reading (WTAR) and reading text at 14 point font

Exclusion Criteria:

* Lack of time and willingness to commit to the completion of this 14-week study
* Less than an 8th grade education
* Having been told by a healthcare provider that they (1) have had a stroke or mini-stroke in the past 12 months, (2) have ever had a traumatic brain injury, (3) have had schizophrenia or psychosis, (4) have problem with alcohol or substance abuse
* extreme difficulty reading ordinary print in a newspaper, or have stopped reading due to poor eyesight.
* extreme difficulty hearing, or being completely unable to hear, ordinary speech in low-noise conditions, even with hearing aid.
* Currently participating in cognitive training or brain training
* Having participated in any cognitive or brain training study within the last 6 months
* Currently participating in yoga or meditation based practices

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline E. Maye, MS, Principal Investigator — University of Florida; Michael Marsiske, PhD, Principal Investigator — University of Florida
Locations (1):
- The Vital Laboratory at the The Village, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared upon request by the study principal investigator. Data to be released will include the variables and participants included in any specific published manuscript, and will be eligible for release twelve months after the date of publication or e-publication in final form.
Time Frame: Data will become available twelve months after the date of publication or e-publication in final form
Access Criteria: All investigators may request data if the request is supported by a research protocol that has been certified as "exempt" by their local Institutional Review Board.

RESULTS

PARTICIPANT FLOW:
Groups:
- Brain Health: Eight weekly group brain health sessions lasting 90-120 minutes. The intervention is psychoeducational, and each week presents information from NIH regarding factors that may promote cognitive health in late life (e.g., sleep, physical activity, social engagement and leisure, cognitive training). Weekly sessions are supplemented with educational videos and group discussion. Weekly homework consists of readings about brain health.
  Participants in both interventions receive all study measures equivalently at all occasions
- Mindfulness-inspired Treatment/Testing: Eight weekly group mindfulness sessions lasting 90-120 minutes, along with a ½ day Mindfulness Retreat at the end of the training period, will include 1) psychoeducation, 2) formal exercises in the form of guided practice mentioned above, and 3) thoughtful exploration of ideas and questions. Formal mindfulness training will follow 21 guided pre-recorded meditative Moving Picture Experts Group Layer-3 Audio (MP3) tracks from the authors for use in class and at home, promoting both fidelity to the model and uniformity in intervention across training groups. Mindfulness activities in the protocol include mindful breathing, eating, walking, and various other practices well documented in the literature to promote mindfulness. Participants will be asked to practice mindfulness on their own time, and to log this.
  Participants receive all of the same measures as the active comparator "Brain Health" condition in Weeks 1-14. In weeks 4-11, participants receive Mindfulness Inspired Treatment
Period: Overall Study
Arm/Group | Brain Health | Mindfulness-inspired Treatment/Testing
Started | 21 | 21
Completed | 19 | 19
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Population: Intent to treat analysis via mixed effects modeling; all available data were used at each occasion. Participants were not able to attend all sessions.
Groups:
- Mindfulness-inspired Treatment/Testing: Eight weekly group mindfulness sessions lasting 90-120 minutes, along with a ½ day Mindfulness Retreat at the end of the training period, will include 1) psychoeducation, 2) formal exercises in the form of guided practice mentioned above, and 3) thoughtful exploration of ideas and questions. Formal mindfulness training will follow 21 guided pre-recorded meditative Moving Picture Experts Group Layer-3 Audio (MP3) tracks from the authors for use in class and at home, promoting both fidelity to the model and uniformity in intervention across training groups. Mindfulness activities in the protocol include mindful breathing, eating, walking, and various other practices well documented in the literature to promote mindfulness. Participants will be asked to practice mindfulness on their own time, and to log this.
  Participants receive all of the same measures as the active comparator "Brain Health" condition in Weeks 1-14. In weeks 4-11, participants receive Mindfulness treatment.
- Total: Total of all reporting groups
Arm/Group | Brain Health | Mindfulness-inspired Treatment/Testing | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.75 (4.83) | 74.95 (6.18) | 73.85 (15.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 21 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 18 | 19 | 37
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Performance in Attention Network Task Conflict Monitoring Over 14 Weekly Measurements
Description: The Attention Network Task is a computerized test that measures three different components of attention (alerting, orienting, and conflict monitoring). Score is the computed as the difference between reaction time on correct trials in cued and uncued conditions. Scores have been normalized via Blom transformation and computed to T-score metric (mean=50, standard deviation = 10, minimum = 0, maximum = 100, higher = worse)
Time Frame: Performance in weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brain Health | Mindfulness-inspired Treatment/Testing
Number analyzed (Participants) | 20 | 20
units on a scale
  Week1: number analyzed (Participants) | 20 | 18
  Week1 | 51.6 (14.4) | 60.4 (8.0)
  Week2: number analyzed (Participants) | 16 | 14
  Week2 | 51.2 (11.7) | 57.3 (10.9)
  Week3: number analyzed (Participants) | 18 | 15
  Week3 | 50.4 (7.6) | 57.1 (7.7)
  Week4: number analyzed (Participants) | 16 | 16
  Week4 | 48.8 (8.3) | 57.9 (9.9)
  Week5: number analyzed (Participants) | 19 | 19
  Week5 | 48.2 (9.8) | 53.8 (10.4)
  Week6: number analyzed (Participants) | 19 | 18
  Week6 | 45.8 (9.8) | 54.4 (9.8)
  Week7: number analyzed (Participants) | 19 | 16
  Week7 | 47.3 (8.5) | 51.7 (9.2)
  Week8: number analyzed (Participants) | 18 | 16
  Week8 | 46.9 (9.7) | 49.2 (9.1)
  Week9: number analyzed (Participants) | 17 | 14
  Week9 | 46.0 (7.9) | 49.7 (8.6)
  Week10: number analyzed (Participants) | 18 | 11
  Week10 | 48.4 (8.1) | 46.7 (8.0)
  Week11: number analyzed (Participants) | 15 | 14
  Week11 | 44.9 (8.3) | 49.7 (8.1)
  Week12: number analyzed (Participants) | 18 | 14
  Week12 | 47.1 (9.4) | 47.3 (8.9)
  Week13: number analyzed (Participants) | 18 | 15
  Week13 | 45.0 (9.4) | 50.4 (8.8)
  Week14: number analyzed (Participants) | 18 | 17
  Week14 | 44.4 (8.9) | 49.2 (7.3)
Statistical Analysis 1: Comparison: Brain Health vs Mindfulness-inspired Treatment/Testing; Mixed effects models were used. Independent variables were linear and quadratic time/occasion, intervention group, and group-by-time interactions if appropriate. Preparatory to modeling, preliminary unconditional models were run to determine best fitting approaches for repeated and random covariance structures. First-order Autoregressive was best (which specifies homogeneous variance over time but allows one correlation between occasions); Test type: Other; p = .024, Mixed Models Analysis — A priori threshold for statistical significance was set at p < .05. No adjustment was made for multiple comparisons. The critical effect of interest evaluated here was the Linear Occasion (1-14) x Group (Brain Health vs. Mindfulness) interaction; F(1,33) = 5.57, p = .024, no adjustments

2. Secondary Outcome: Performance in Useful Field of View Over 14 Weekly Measurements
Description: The useful field of view task is a computer-administered selective visual attention test that determines the minimum presentation time needed (between 16-500 msec) to correctly make two visual judgments: (a) is a centrally presented line drawing of a car or truck? and (b) where on the screen is a peripheral car located? Score is the fastest presentation time at which participants achieve at least 75% accuracy. Scores have been normalized via Blom transformation and computed to T-score metric (mean=50, standard deviation = 10, minimum = 0, maximum = 100, higher = worse)
Time Frame: Performance in weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brain Health | Mindfulness-inspired Treatment/Testing
Number analyzed (Participants) | 20 | 20
units on a scale
  Week1: number analyzed (Participants) | 18 | 20
  Week1 | 52.3 (8.4) | 57.0 (8.3)
  Week2: number analyzed (Participants) | 15 | 15
  Week2 | 52.9 (10.0) | 53.7 (8.0)
  Week3: number analyzed (Participants) | 17 | 14
  Week3 | 52.1 (9.4) | 53.9 (11.8)
  Week4: number analyzed (Participants) | 16 | 16
  Week4 | 52.2 (9.0) | 51.3 (8.6)
  Week5: number analyzed (Participants) | 17 | 18
  Week5 | 49.7 (9.1) | 55.1 (9.6)
  Week6: number analyzed (Participants) | 18 | 18
  Week6 | 47.9 (8.0) | 51.4 (8.2)
  Week7: number analyzed (Participants) | 17 | 15
  Week7 | 46.1 (9.3) | 47.8 (7.4)
  Week8: number analyzed (Participants) | 17 | 16
  Week8 | 49.9 (9.6) | 49.5 (8.4)
  Week9: number analyzed (Participants) | 16 | 13
  Week9 | 49.8 (9.6) | 46.9 (9.4)
  Week10: number analyzed (Participants) | 17 | 11
  Week10 | 50.5 (9.1) | 45.7 (9.2)
  Week11: number analyzed (Participants) | 14 | 13
  Week11 | 45.3 (9.1) | 49.2 (10.4)
  Week12: number analyzed (Participants) | 17 | 14
  Week12 | 48.8 (13.3) | 45.3 (7.6)
  Week13: number analyzed (Participants) | 17 | 14
  Week13 | 47.9 (11.2) | 46.0 (8.2)
  Week14: number analyzed (Participants) | 18 | 16
  Week14 | 48.1 (11.5) | 47.2 (9.4)
Statistical Analysis 1: Comparison: Brain Health vs Mindfulness-inspired Treatment/Testing; Mixed effects models were used. Independent variables were linear and quadratic time/occasion, intervention group, and group-by-time interactions if appropriate. Preparatory to modeling, preliminary unconditional models were run to determine best fitting approaches for repeated and random covariance structures. Diagonal repeated covariance was best (heterogeneous variance over time, and no residual cross-time covariances); Test type: Other; p = 0.333, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F(1,34) = 0.96, p = .333, no adjustments

3. Secondary Outcome: Performance in Stroop Interference Over 14 Weekly Measurements
Description: This task set is computerized presents participants with a word (red or green or blue) that may be presented in (a) congruent (same) color as the word itself (e.g., red word is printed in red), or (b) incongruent (word red printed in green or blue). Participants are cued to either select the word or the color, this varies from trial to trial. Score is the reaction time difference between correct responses to congruent and incongruent stimuli. Scores have been normalized via Blom transformation and computed to T-score metric (mean=50, standard deviation = 10, minimum = 0, maximum = 100, higher = worse)
Time Frame: Performance in weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brain Health | Mindfulness-inspired Treatment/Testing
Number analyzed (Participants) | 20 | 20
units on a scale
  Week1: number analyzed (Participants) | 20 | 19
  Week1 | 51.5 (8.6) | 54.7 (9.0)
  Week2: number analyzed (Participants) | 16 | 13
  Week2 | 53.6 (8.4) | 49.5 (12.0)
  Week3: number analyzed (Participants) | 18 | 14
  Week3 | 50.8 (11.0) | 49.2 (12.1)
  Week4: number analyzed (Participants) | 16 | 16
  Week4 | 52.9 (10.1) | 51.3 (11.4)
  Week5: number analyzed (Participants) | 17 | 18
  Week5 | 50.7 (8.9) | 50.0 (10.2)
  Week6: number analyzed (Participants) | 18 | 18
  Week6 | 50.9 (9.1) | 51.0 (8.2)
  Week7: number analyzed (Participants) | 18 | 15
  Week7 | 49.8 (8.1) | 50.0 (13.1)
  Week8: number analyzed (Participants) | 18 | 16
  Week8 | 49.5 (9.8) | 49.0 (7.9)
  Week9: number analyzed (Participants) | 17 | 13
  Week9 | 47.3 (10.5) | 51.6 (9.5)
  Week10: number analyzed (Participants) | 18 | 11
  Week10 | 49.4 (9.2) | 45.8 (8.8)
  Week11: number analyzed (Participants) | 15 | 14
  Week11 | 50.9 (12.5) | 50.0 (10.1)
  Week12: number analyzed (Participants) | 17 | 14
  Week12 | 47.0 (8.9) | 45.1 (7.3)
  Week13: number analyzed (Participants) | 18 | 15
  Week13 | 48.9 (10.8) | 51.1 (9.2)
  Week14: number analyzed (Participants) | 18 | 17
  Week14 | 48.9 (12.8) | 47.8 (11.4)

4. Other Pre Specified Outcome: Self-ratings of Perceived Mind Wandering Over 8 Weekly Measurements
Description: Participants in both arms are asked, at the end of each of their eight intervention sessions, to focus on breathing. They are interrupted five times during this breathing exercise and asked what proportion of their attention (0-100) was wandering off the breathing task. Score is the average proportion of self-rated mind-wandering over five probes. Scores have been normalized via Blom transformation and computed to T-score metric (mean=50, standard deviation = 10, minimum = 0, maximum = 100, higher = worse)
Time Frame: Self-ratings of weeks 4, 5, 6, 7, 8, 9, 10, 11
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brain Health | Mindfulness-inspired Treatment/Testing
Number analyzed (Participants) | 20 | 20
units on a scale
  Week4: number analyzed (Participants) | 18 | 18
  Week4 | 50.5 (7.9) | 54.3 (10.3)
  Week5: number analyzed (Participants) | 19 | 19
  Week5 | 50.6 (7.7) | 51.7 (9.6)
  Week6: number analyzed (Participants) | 20 | 19
  Week6 | 51.1 (9.5) | 52.5 (10.4)
  Week7: number analyzed (Participants) | 20 | 18
  Week7 | 50.7 (11.5) | 49.7 (10.2)
  Week8: number analyzed (Participants) | 19 | 18
  Week8 | 51.2 (10.3) | 51.4 (12.1)
  Week9: number analyzed (Participants) | 16 | 15
  Week9 | 50.9 (10.7) | 47.5 (10.1)
  Week10: number analyzed (Participants) | 16 | 13
  Week10 | 48.9 (9.7) | 44.9 (9.3)
  Week11: number analyzed (Participants) | 14 | 15
  Week11 | 46.0 (7.7) | 44.2 (8.7)
Statistical Analysis 1: Comparison: Brain Health vs Mindfulness-inspired Treatment/Testing; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.001, Mixed Models Analysis — A priori threshold for statistical significance was set at p < .05. No adjustment was made for multiple comparisons. The critical effect of interest evaluated here was the Linear Occasion (1-8) x Group (Brain Health vs. Mindfulness) interaction; F(1,31.069) = 15.046, p = .001, no adjustments

5. Other Pre Specified Outcome: Self-ratings in Anxiety (GAD-7) Questionnaire Over 14 Weekly Measurements
Description: Participants will answer computer 7 administered questions about anxiety in the past week. Score is a Likert-type scale response from the following scale: 0=not at all, 1=several days, 2=more than half the days, 3=nearly every day. Scores have been normalized via Blom transformation and computed to T-score metric (mean=50, standard deviation = 10, minimum = 0, maximum = 100, higher = worse)
Time Frame: Self-ratings in weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brain Health | Mindfulness-inspired Treatment/Testing
Number analyzed (Participants) | 20 | 20
units on a scale
  Week1 | 50.5 (7.6) | 53.5 (10.0)
  Week2: number analyzed (Participants) | 16 | 15
  Week2 | 51.3 (10.9) | 50.4 (6.7)
  Week3: number analyzed (Participants) | 18 | 15
  Week3 | 50.2 (10.1) | 53.0 (8.4)
  Week4: number analyzed (Participants) | 16 | 15
  Week4 | 47.8 (9.3) | 51.8 (9.6)
  Week5: number analyzed (Participants) | 18 | 19
  Week5 | 50.3 (9.6) | 52.5 (8.3)
  Week6: number analyzed (Participants) | 19 | 19
  Week6 | 59.2 (7.8) | 51.8 (8.4)
  Week7: number analyzed (Participants) | 18 | 16
  Week7 | 49.0 (7.8) | 50.0 (9.2)
  Week8: number analyzed (Participants) | 15 | 16
  Week8 | 49.2 (8.2) | 49.0 (8.2)
  Week9: number analyzed (Participants) | 17 | 13
  Week9 | 52.0 (10.5) | 49.3 (8.9)
  Week10: number analyzed (Participants) | 17 | 11
  Week10 | 50.3 (9.4) | 50.4 (7.2)
  Week11: number analyzed (Participants) | 15 | 14
  Week11 | 51.2 (9.9) | 50.5 (10.8)
  Week12: number analyzed (Participants) | 17 | 14
  Week12 | 50.0 (9.2) | 50 (10)
  Week13: number analyzed (Participants) | 18 | 15
  Week13 | 50.7 (10.7) | 49.1 (9.9)
  Week14: number analyzed (Participants) | 18 | 17
  Week14 | 48.5 (8.0) | 49.9 (8.3)
Statistical Analysis 1: Comparison: Brain Health vs Mindfulness-inspired Treatment/Testing; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.448, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F(1,34) = 0.589, p = .0.448, no adjustments

6. Other Pre Specified Outcome: Self-ratings on Cognitive and Affective Mindfulness Scale (CAMSr) Over 14 Weekly Measurements
Description: Cognitive and Affective Mindfulness Scale (CAMSr) will be computer administered. It is a psychological measurement to explore mindfulness. Each week ten items are rated on a 4-point Likert-type scale (1=rarely/never, 2=sometimes, 3=often, 4=almost always). Higher scores indicate greater cognitive and emotional focus. Scores are the average of the ten items, normalized and converted to T-score (mean=50, standard deviation = 10, minimum = 0, maximum = 100, higher = better) metric.
Time Frame: Self-ratings weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brain Health | Mindfulness-inspired Treatment/Testing
Number analyzed (Participants) | 20 | 20
units on a scale
  Week1: number analyzed (Participants) | 19 | 20
  Week1 | 48.8 (8.3) | 48.8 (8.5)
  Week2: number analyzed (Participants) | 16 | 15
  Week2 | 49.4 (9.9) | 50.3 (8.8)
  Week3: number analyzed (Participants) | 18 | 15
  Week3 | 49.9 (10.9) | 47.7 (7.6)
  Week4: number analyzed (Participants) | 15 | 16
  Week4 | 53.3 (9.3) | 46.0 (10.1)
  Week5: number analyzed (Participants) | 18 | 18
  Week5 | 51.3 (11.6) | 47.0 (8.8)
  Week6: number analyzed (Participants) | 19 | 18
  Week6 | 51.2 (7.8) | 48.6 (8.5)
  Week7: number analyzed (Participants) | 18 | 15
  Week7 | 50.7 (9.7) | 49.7 (9.4)
  Week8: number analyzed (Participants) | 17 | 16
  Week8 | 49.0 (11.1) | 50.3 (10.2)
  Week9: number analyzed (Participants) | 15 | 12
  Week9 | 50.0 (11.0) | 47.9 (11.0)
  Week10: number analyzed (Participants) | 18 | 11
  Week10 | 50.3 (8.8) | 49.7 (11.6)
  Week11: number analyzed (Participants) | 14 | 13
  Week11 | 51.8 (10.0) | 48.7 (13.2)
  Week12: number analyzed (Participants) | 17 | 14
  Week12 | 50.9 (9.3) | 48.5 (9.6)
  Week13: number analyzed (Participants) | 18 | 15
  Week13 | 51.6 (8.8) | 51.4 (9.0)
  Week14: number analyzed (Participants) | 19 | 15
  Week14 | 51.4 (10) | 51.3 (10.6)
Statistical Analysis 1: Comparison: Brain Health vs Mindfulness-inspired Treatment/Testing; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.439, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; F(1,31) = 0.616, p = 0.439, no adjustments

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the period of each participant's participation, 14 weeks.
Arm/Group | Brain Health | Mindfulness-inspired Treatment/Testing
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT02714426/Prot_SAP_000.pdf